CLINICAL TRIAL: NCT02262208
Title: Exercise as a Tool for Studying the Mechanisms and Applicability of Glycemic Variability in Individuals With and Without Type 2 Diabetes Mellitus
Brief Title: Exercise as a Tool for Studying the Mechanisms and Applicability of Glycemic Variability
Acronym: ETSMAGV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Beatriz D'Agord Schaan, Beatriz D'Agord Schaan, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 120148
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
Keywords: Glycemic variability, exercise, diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus | interventions — Exercise; Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with type 2 diabetes (Other)
  Interventions: Other: Aerobic Exercises; Other: Eccentric Exercise; Device: Continuous glucose monitoring system (Guardian, Medtronic, Northridge, USA)
- Healthy (Other)
  Interventions: Other: Aerobic Exercises; Other: Eccentric Exercise; Device: Continuous glucose monitoring system (Guardian, Medtronic, Northridge, USA)

INTERVENTIONS:
Other: Aerobic Exercises — Exercise intensity for each individual by a heart rate monitor (Polar F1 TM, Polar Electro Oy, Helsinki, Finland), and a Borg 0-10 scale used to register individuals' perceived exertion every 5 minutes throughout the experimental sessions.
  Aerobic session will consist of 40 min of lower limb bicycle at 70% of the peak heart rate, as determined in the incremental exercise test.
Other: Eccentric Exercise — Eccentric session will consist of 40 min of one lower -limb exercises (leg press) with 6 sets of 10 repetitions at 120% of 1-RM.
Device: Continuous glucose monitoring system (Guardian, Medtronic, Northridge, USA) — Subjects will be admitted to the laboratory in the morning at approximately 9:00 a.m., 24 h before the exercise session, when the glucose sensor (Sof-SensorTM, Medtronic Mini-Med, Northridge, USA) will be inserted subcutaneously. The sensor is a glucose oxidase based platinum electrode that is inserted through a needle into the subcutaneous tissue of the anterior abdominal wall, using a spring-loaded device (Senserter, Medtronic, Northridge, USA). Glucose profiles will be collected the day before (day 1), the day of (day 2), and the day following (day 3) and 40 min of exercise. Each sensor will be used continuously for up to 72 h.

SUMMARY:
The aim this study is characterize glycemic variability using linear and nonlinear mathematical tools, under basal conditions and in response to specific protocols acute exercise that evoke oxidative stress and inflammation in healthy subjects and type 2 diabetes patients. For this purpose, the sample size will consist of 37 individuals healthy and 32 without type 2 diabetes mellitus wore a CGMS during 3 days. Participants randomly performed aerobic and eccentric sessions, both in the morning (24h after CGMS placement), and at least 7 days apart. Glucose variability was evaluated by glucose standard deviation, glucose variance, mean amplitude of glycemic excursions (MAGE), and glucose coefficient of variation (conventional methods) as well as by spectral and symbolic analysis (non-conventional methods). Physiological mechanisms altered by exercise protocols (Human Soluble Interleukin-6 and Glutathione), will be measured in blood samples.

DETAILED DESCRIPTION:
The aim this study is characterize glycemic variability using linear and nonlinear mathematical tools, under basal conditions and in response to specific protocols acute exercise that evoke oxidative stress and inflammation in healthy subjects and type 2 diabetes patients. For this purpose, the sample size will consist of 37 individuals healthy and 32 without type 2 diabetes mellitus, which will undertake the two types of exercise, randomly distributed. The maximal incremental exercise test will be performed in electrically braked cycle ergometer (ER-900, Jaeger, Wu¨ rzburg, Germany) in order to assess possible contraindications to the proposed protocol as well functional capacity, which will be used in prescription of the aerobic exercise session and a testing strength maximal will be conducted and used in the prescription of the eccentric exercise session.

The glucose variability will be assessed by continuous glucose monitoring system (CGMS) during 72h. Glucose variability will be evaluated by glucose standard deviation, glucose variance, mean amplitude of glycemic excursions (MAGE), and glucose coefficient of variation (conventional methods) as well as by spectral and symbolic analysis (non-conventional methods). Physiological mechanisms altered by exercise protocols will be measured in blood samples., Human Soluble Interleukin-6 ( HU IL 6 ELISA KIT - BIOSOURCE) and Glutathione (GSH) indicator of oxidative stress (GSH assay in: Rahman I, Kode A, Biswas SK. Nat Protoc. 2006;1(6):3159-65). The aerobic session will consist of 40 min of lower limb bicycle at 70% of the peak heart rate, as determined in the incremental exercise test and eccentric session will consist of 40 min of one lower -limb exercises (leg press) with 6 sets of 10 repetitions at 120% of 1-RM. The protocol was approved by the Ethics in Research Committee at Hospital de Clínicas de Porto Alegre and all patients will provide their written informed consent before the participation.The research will be performed at the Exercise Pathophysiology Research laboratory of the Hospital de Clínicas de Porto Alegre. We believe that signs of glycemic variability has characteristics detectable by alternative, related to hysiological processes such as oxidative stress and inflammation, evoked by aerobic and eccentric exercise protocols mathematical methods, may help explain the acute response of healthy individuals and patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes Male and female 18-65 years old

Exclusion Criteria:

Chronic kidney failure; Limb amputation Diabetic proliferative retinopathy; Regular physical training; Severe autonomic neuropathy; Diabetic nephropathy established; Coronary artery disease; Heart failure; Uncontrolled hypertension Treatment of insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability by continuous glucose monitoring system | The monitor that analyzes the data every 10s and reports average values every 5 min, totalizing 288 readings per day. Glucose profiles will be collected the day before (day 1), the day of (day 2), and the day following (day 3) of 40 min of both exercise.
  Will be assessed conventional and non-conventional methods to analyze glucose variability derived from multiple measurements performed with continuous glucose monitoring system (CGMS).Subjects will be admitted to the laboratory in the morning at approximately 9:00 a.m., 24 h before the exercise session, when the glucose sensor (Sof-SensorTM, Medtronic Mini-Med, Northridge, USA) will be inserted subcutaneously. The sensor is a glucose oxidase based platinum electrode that is inserted through a needle into the subcutaneous tissue of the anterior abdominal wall, using a spring-loaded device (Senserter, Medtronic, Northridge, USA). Glucose profiles will be collected the day before (day 1), the day of (day 2), and the day following (day 3) and 40 min of exercise. Each sensor will be used continuously for up to 72 h.

SECONDARY OUTCOMES:
Oxidative stress | 10 minutes before the exercise sessions and 10 minutes after the exercise sessions.
  Will be assessed by Glutathione (GSH) indicator of oxidative stress (GSH assay in: Rahman I, Kode A, Biswas SK Nat PROTOC 2006, 1 (6): 3159-65.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Rahman I, Kode A, Biswas SK. Assay for quantitative determination of glutathione and glutathione disulfide levels using enzymatic recycling method. Nat Protoc. 2006;1(6):3159-65. doi: 10.1038/nprot.2006.378. PMID 17406579
- [Derived] Figueira FR, Umpierre D, Bock PM, Waclawovsky G, Guerra AP, Donelli A, Andrades M, Casali KR, Schaan BD. Effect of exercise on glucose variability in healthy subjects: randomized crossover trial. Biol Sport. 2019 Jun;36(2):141-148. doi: 10.5114/biolsport.2019.83006. Epub 2019 Feb 22. PMID 31223191